CLINICAL TRIAL: NCT04233398
Title: A Multi-center, Randomized, Controlled Trial of High Intensity Focused Ultrasound (HIFU) Treatment of Benign Thyroid Nodules
Brief Title: HIFU Treatment of Benign Thyroid Nodules
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIFU20190725
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Nodule (Benign)
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: Patients in the test group will be treated with high intensity focused ultrasound (HIFU), while patients in the control group will be actively observed and followed up by ultrasound examination. during the follow-up period, the follow-up visits time and follow-up examination items (clinical examination, ultrasonic examination and laboratory examination etc.) were the same in the both groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group HIFU treatment (Experimental): Patients in the test group (120) will be treated with high intensity focused ultrasound (HIFU). The primary objective of this clinical trial is to evaluate the efficacy of the test device in the treatment of benign thyroid nodules, and the secondary objective is to evaluate the safety of the test device in the treatment of benign thyroid nodules and the improvement of symptoms (VAS score).
  Interventions: Device: Device: Echopulse (HIFU ablation)
- Control group (No Intervention): Patients in the control group (120) will be actively observed and followed up. The primary objective of this clinical trial is to evaluate the efficacy of the test device in the treatment of benign thyroid nodules, and the secondary objective is to evaluate the safety of the test device in the treatment of benign thyroid nodules and the improvement of symptoms (VAS score).

INTERVENTIONS:
Device: Device: Echopulse (HIFU ablation) — High-intensity focused ultrasound (HIFU) is a non-invasive, non-invasive treatment method. The principle is to focus high-intensity ultrasound on the target area. Energy is absorbed by the target tissue and converted into thermal energy. The local temperature quickly reaches a maximum of 85 ° C. It induces coagulative necrosis of focus tissue cells, but does not damage the tissues surrounding the treatment targ
  Arms: Test group HIFU treatment

SUMMARY:
This clinical trial is to evaluate the effectiveness and the safety of high intensity focused ultrasound (HIFU) in the treatment of benign thyroid nodules.

DETAILED DESCRIPTION:
This clinical trial is a prospective, multicentre, randomized, controlled study of high intensity focused ultrasound (HIFU) treatment of benign thyroid nodules. this study will include 240 patients with benign thyroid nodules that meet all ths the inclusion / exclusion criteria and will be randomly divided into two groups at 1: 1 ratio. Patients in the test group will be treated with high intensity focused ultrasound (HIFU), while patients in the control group will be actively observed and followed up by ultrasound examination. The primary objective of this clinical trial is to evaluate the efficacy of the test device in the treatment of benign thyroid nodules, and the secondary objective is to evaluate the safety of the test device in the treatment of benign thyroid nodules and the improvement of symptoms assessed by VAS score.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients older than 18 years and younger than 70 years
2. No history of neck irradiation
3. Normal thyroid function, serum calcitonin level, PTH and serum calcium at screening visit examination.
4. No abnormal cervical lymph nodes during screening visit examination.
5. The target thyroid nodule must meet all of the following conditions:

   1. Single nodule, 2cm≤max diameter≤4cm
   2. Causing appearance , pressure or swallowing symptoms
   3. Composition of target nodule: solid or predominantly solid (solid area≥80%)
   4. Ultrasound imaging of target nodule assessed by 2017 ACR TI-RADS(≤Grade 3), and proved benign by once FNA (bethesda categoryⅡ); Ultrasound imaging of target nodule assessed by 2017 ACR TI-RADS( Grade 4), and proved benign by twice FNA (bethesda categoryⅡ).
   5. The distance from the posterior edge of the target nodule to the skin is not less than 12.3mm, and the depth from the anterior edge of the target nodule to the skin is not more than 19.4mm.
   6. No macro-calcifications in target nodule, macro-calcifications induce a significant shadow in the ultrsound imaging.
   7. the skin is free from any significant thick scars.
6. If there are more than one nodule on the treatment side, all of the following conditions shall be met:

   1. No more than 2 nodules except the target nodule.
   2. Maximum diameter of the nodules is smaller than 1 cm and ultrasound imaging ≤ Grade 3 assessed by 2017 ACR TI-RADS.
7. If there are nodules on the opposite side of HIFU treatment side, one of the following conditions shall be met:

   1. Maximum diameter of these nodules is smaller than 1 cm and ultrasound imaging ≤ Grade 3 assessed by 2017 ACR TI-RADS.
   2. Only one nodule with 1cm≤ max diameter < 2cm, or/and no more than three nodule with max diameter <1cm. Ultrasonic images of all nodules≤Grade 3 assessed by 2017 ACR TI-RADS.
8. Absence of abnormal vocal cord mobility at laryngoscopy.
9. Patients reject or cannot tolerate invasive surgical treatment.
10. Patient has signed a written informed consent.

Exclusion Criteria:

1. The ultrasound report indicated that follicular tumors were not excluded.
2. Known history of thyroid cancer or other neoplasias in the neck region.
3. Head and/or neck disease that prevents hyper-extension of neck.
4. Patients currently in the acute phase of any disease.
5. History of head and neck, pulmonary and systemic infections in the last 2 weeks.
6. The white blood cell test result exceeded the upper limit of the normal range.
7. Tenderness of the thyroid and/or thyroid nodules.
8. History of arrhythmia, coronary heart disease or valvular heart disease, heart failure.
9. The blood pressure is not controlled after the combination of three antihypertensive drugs (SBP ≥ 140 mmHg, DBP ≥ 90 mmHg)
10. COPD history or acute phase of asthma attach
11. Patients with liver dysfunction ( ALT or AST level 2.5 times higher than the upper limit of the normal reference range)
12. Patients with renal insufficiency( eGFR< 45ml/min/1.73m2).
13. Fasting blood glucose >8mmol/L after hypoglycemic drug treatment
14. Patients currently sufferrign from hematological diseases or bleeding tendency, or patients currently requiring continuous administration of antiplatelet and anticoagulant drugs
15. Pregnant or lactating woman
16. Woman who Plan to be pregnant during the study period.
17. Any contraindication to the assigned analgesia/ anaesthesia.
18. Patients who participated in other clinical trials in the past 3 months.
19. Alzhemier's patients or patient with cognitive impairment.
20. Other patients judged by the investigators to be unsuitable for the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Effectiveness evaluation using treatment effective rate | 12 Months
  percentage of patients who achieve treatment success (volume reduction ratio > 50%) at 12 months after HIFU treatment assessed by ultrasound examination

SECONDARY OUTCOMES:
Symptoms score improvement | 12 Months
  Using Visual Analogic Scale between (0-100 mm) to evaluate the improvement of appearance symptoms, compression symptoms and swallowing symptoms and pain.
  With 0 being no pain and 100 being the worst pain imaginable
Incidence of Treatment-Emergent Adverse Events | 12 Months
  Incidence of local and/or general adverse reactions and other related symptoms at 1, 7 days and 1, 3, 6 and 12 months follow-up after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kuang, MD, Principal Investigator — Guangdong Province People's Hopital

IPD SHARING:
Plan to Share IPD: No